CLINICAL TRIAL: NCT05130489
Title: Chimeric Antigen Receptor (CAR) Cell Therapy Related Cardiovascular Outcomes
Brief Title: CAR T Cell Therapy Related Cardiovascular Outcomes
Acronym: CARTCO
Status: Completed | Type: Observational
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Derek Yellon, Professor, University College London Hospitals
Other Study IDs: 20/SC/0301
Record Dates: First submitted 2021-11-04; First posted 2021-11-23 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Diseases; B-cell Acute Lymphoblastic Leukemia; B-cell Lymphoma Refractory; B-cell Lymphoma Recurrent; Primary Mediastinal Large B-cell Lymphoma (PMBCL); Diffuse Large B Cell Lymphoma; Cardiotoxicity; Cardiovascular Complication
Keywords: Cardio-oncology; CAR T cell therapy; Cardiotoxicity
MeSH Terms: conditions — Cardiovascular Diseases; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum will be separated from whole blood and retained for follow-on analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This will be a cohort study of all patients receiving Cluster of Differentiation 19 (CD19)-specific CAR T cell therapy for relapsed/refractory B cell haematological malignancies. Patients will receive cardiac assessment and have serum cardiac biomarkers, ECG, transthoracic echocardiogram and cardiac magnetic resonance imaging performed at baseline prior to CAR T cell therapy, 7 days post CAR T cell infusion, and 3 months post CAR T cell infusion. Abnormalities in these cardiac investigations will be used to demonstrate cardiac injury and identify which patients are most at risk of developing cardiac injury related to CAR T cell therapy.

DETAILED DESCRIPTION:
CD19-specific chimeric antigen receptor (CAR) T cells are a novel therapy for relapsing or refractory blood cancers, which have delivered a significant improvement in the rates of complete and partial remission. However, they are associated with toxicities, with some of early evidence suggestive of cardiovascular involvement. Despite this, the full extent of cardiovascular toxicity is poorly understood.

This research study seeks to understand the cardiac safety of CAR T cells in patients who receive this therapy as part of standard care for relapsed/refractory B-cell blood cancer. They will be assessed for cardiovascular risk factors via history, blood biomarkers, and cardiac imaging tests. These parameters will be repeated at 7 days following administration of the CAR T cells or if there are signs of cardiovascular deterioration, and again at 3 months follow up.

The aim is to predict the cohort most at risk of cardiovascular toxicity, and demonstrate evidence of cardiac injury on the cardiac imaging scans.

ELIGIBILITY:
Inclusion Criteria:

* Patients with capacity, (aged 16 and older)
* Undergoing CAR T cells for treatment for relapsing or refractory haematological malignancies

Exclusion Criteria:

* Patients under 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving CD19-specific CAR T cell therapy for the management of relapsing or refractory haematological malignancy at the MacMillan Cancer Centre within the University College London Hospital will be considered for participation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Detected abnormalities - Composite | 3 months
  The primary outcome is a composite of detected abnormalities on biomarkers, transthoracic echocardiogram (TTE), or Cardiac magnetic resonance (CMR) following CAR T cell infusion.

SECONDARY OUTCOMES:
Detected abnormalities - Individual | 3 months
  The secondary outcome measures includes a composite of detected abnormalities of factors on cardiac biomarkers (troponin and N-terminal pro B-type natriuretic peptide) , electrocardiogram (ECG) changes and acute heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No